CLINICAL TRIAL: NCT02727673
Title: A Prospective Randomized Trial on the Relationship Between Circulating Tumor Stem Cells and the Clinical Pathology
Brief Title: Relationship Between Circulating Tumor Stem Cells and the Clinical Pathology
Status: Completed | Type: Observational
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Other Study IDs: ZD201200102-P1
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Cancer Stem Cells; Postoperative Recurrence and Metastasis; Hepatocellular Carcinoma
Keywords: cancer stem cells
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- healthy volunteers: matched group
- hepatitis cirrhosis: negative group
- hepatocellular carcinoma: patients with primary HCC

SUMMARY:
The aim of this study is to establish a platform of detecting and sorting circulating tumor stem cells from peripheral blood in HCC patients; to investigate the relationship between circulating tumor stem cells and their effects on postoperative recurrence and metastasis, in order to provide a new therapeutic target for hepatocellular carcinoma treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years and <=70 years of age;
2. No dysfunction in major organs; Blood routine, kidney function, cardiac function and lung function are basically normal.
3. Patients who can understand this trial and have signed information consent

Exclusion Criteria:

1. Reject to attend；
2. Impossible to come to our hospital for physical examination regularly;
3. Patients with other diseases which may affect the treatment mentioned

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 250 healthy volunteers, 250 patients with hepatitis cirrhosis, 500 patients with HCC;
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the overall survival rate of each group | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China